CLINICAL TRIAL: NCT00172146
Title: Influences of Cane Use on Voluntary Forward Stepping Movement and Associated Attentional Demands in Hemiplegic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361700329
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Stroke
Keywords: Hemiplegia; Regular cane; Volitional stepping; Dynamic equilibrium; Attention; Dual task
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The purpose of this study was to examine the influence of cane use on the movement, kinetics, and associated attentional demands of performing a voluntary forward stepping movement in patients with stroke and age-matched healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Age ang Sex are correspond with the stroke subjects(between 30 and 75 years old)
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital

Stroke subjects

* between 30 and 75 years old
* stroke confirmed by ICD-10-CM (including I60, I61, I62, I63, I67, and I63.9)
* first stroke with single side hemiplegia and received acute treatment at NTUH
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital
* able to stand independently for 10 minutes and to forward step without ankle-foot orthosis
* Mini-Mental State Examination (MMSE) score at least 24

Excursion criteria:

Healthy subjects

* having other neurological diseases, or moderate to severe neuromuscular or musculoskeletal disorders, or disorders from systematic diseases those would influence the belance or motor ability

Stroke subjects

* having unstable vital sign, unconsciousness, or obvious cognitive, perception, and language impairment, and couldn't communicate with the experimenters
* having other neurological diseases, or moderate to severe neuromuscular or musculoskeletal or cardiovascular disorders, or disorders from systematic diseases those will influence standing ability other than stroke
* having hemi-neglect or hemi-anopia

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2002-08; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Province of China, Taiwan